CLINICAL TRIAL: NCT06522685
Title: Neural and Immune Correlates of Painful Chemotherapy-Induced Neuropathy, Feasibility and Preliminary Efficacy of a Motor Cortex Non-Invasive Brain Stimulation Intervention
Brief Title: Neural and Immune Correlates of CIPN and Possible Analgesic Effect of Non-invasive Motor Cortex Stimulation
Acronym: NIBS4CIPN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morgan State University (Other)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: HP-00111489
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chronic Pain; Neuropathy; Neuropathic Pain; Non-invasive brain stimulation; transcranial direct current stimulation
MeSH Terms: conditions — Chronic Pain; Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double-Blind Sham-controlled Parallel comparing feasibility in non-Hispanic black participants to non-Hispanic white participants (2 arms, 2 groups each arm; total 4 groups with 20 participants in a group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A numerical code will be put into the device by the participant which will determine whether the device is in real or sham mode. The principal investigator, evaluator and al study staff excepting the device company and study statistician will be blinded to this code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Left motor cortex targeted anodal transcranial direct current stimulation (Experimental): Active left motor cortex targeted anodal transcranial direct current stimulation at 2 milliamperes applied for 20 minutes once daily on Monday through Friday for two consecutive weeks.
  Interventions: Device: transcranial direct current stimulation Soterix REMOTE 1x1 miniCT
- Left motor cortex targeted sham transcranial direct current stimulation (Sham Comparator): Active left motor cortex targeted anodal transcranial direct current stimulation at 0 milliamperes applied for 20 minutes once daily on Monday through Friday for two consecutive weeks. The sham consists of a ramp up to 2 mA and immediate ramp down to 0 mA at the beginning of the 20 minute period and a ramp up to 2 mA and immediate ramp down to 0 mA at the end of the 20 minute period.
  Interventions: Device: transcranial direct current stimulation Soterix REMOTE 1x1 miniCT

INTERVENTIONS:
Device: transcranial direct current stimulation Soterix REMOTE 1x1 miniCT — Soterix Medical REMOTE Neuromodulation is the only system with device, accessories, and software designed for deployed use. Safe transcranial Electrical Stimulation requires advanced systems designed for consistency and control. REMOTE Neuromodulation is the only system designed from the ground up to allow translation of clinical tES, including tDCS protocols, to diverse deployed environments, while maintaining medical standards.
  Other Names: tDCS; Soterix REMOTE 1x1 miniCT

SUMMARY:
Over half of cancer patients receiving common chemotherapy treatments experience painful nerve damage called chemotherapy-induced peripheral neuropathy (CIPN). Non-Hispanic Black (NHB) patients are more likely to suffer from this condition and more often need to reduce their chemotherapy doses compared to Non-Hispanic White (NHW) patients.

Currently, only one medication, duloxetine, is approved for treating CIPN, but it doesn't work for everyone. A new approach, transcranial direct current stimulation (tDCS), shows promise as a safe and effective treatment. tDCS can be done at home and reduces the need for hospital visits.

Research indicates that tDCS can improve pain responses in the brain's pain control network. There are differences in pain sensitivity and brain activity related to pain between NHB and NHW individuals, which may influence the effectiveness of treatments.

This research aims to conduct a study to:

1. Test if tDCS is a helpful treatment for painful CIPN.
2. Investigate how CIPN affects brain function in NHB and NHW patients.
3. Examine the role of inflammation in CIPN and its connection to pain severity and brain function.

The investigators expect that NHB patients will benefit more from tDCS due to differences in their brain's pain response system. This project aims to address health disparities and improve outcomes for urban communities, particularly in Baltimore.

DETAILED DESCRIPTION:
More than half of patients treated with commonly used platinum- and taxane-based anti-cancer agents suffer painful chemotherapy-induced peripheral neuropathy (CIPN). Non-Hispanic Black (NHB) patients have a greater risk (risk ratio=1.6-2.4) of experiencing clinically relevant CIPN and consequent chemotherapy dose reductions compared to non-Hispanic Whites (NHWs). Despite the greater risk of painful CIPN in NHB cancer patients, clinical trials in patients suffering with CIPN have historically included homogeneous patient populations of NHWs. Only duloxetine is approved to treat painful CIPN and is not effective for or tolerated by all patients. Transcranial direct current stimulation (tDCS) of the motor cortex is emerging as a promising, safe, and effective intervention for the pain of neuropathy. An additional benefit of tDCS is that it can be administered at home and supervised remotely, minimizing stressful visits to a hospital venue for treatment. A recent randomized experimental study in healthy individuals completed by the PI showed that one 20-minute session of motor cortex tDCS reduced capsaicin-induced hyperalgesia. To understand the mechanism of pain ameliorating effects of motor cortex tDCS, the PI found enhanced neurophysiological responses of the descending pain modulatory network (DPMN), a group of brain structures activated in response to painful stimuli, after active compared to sham stimulation. Previous investigations have observed differences in opioid receptor binding and pain responses in the DPMN (notably the cingulate cortex and ventral striatum) between healthy NHBs and NHWs as well as differences in pain sensitivity. Likely relevant to the mechanism of CIPN, PET scanning of chemotherapy patients reveals neuroinflammation throughout the brain. The facts that 1) NHB individuals experience a greater rate of CIPN, but have not been represented in relevant clinical studies, 2) non-invasive tDCS is emerging as a safe and effective treatment for neuropathic pain and can be implemented in the home 3) the DPMN is implicated in central pain responses and is activity is enhanced after tDCS and 4) neuroinflammation likely plays a role in CIPN have led us to the present research plan. The overarching goal of this proposal to conduct an exploratory double-blind randomized controlled trial (RCT) addressing 3 specific aims: 1) determine the feasibility and efficacy of active tDCS targeting motor cortex as an analgesic and antihyperalgesic intervention in patients with painful CIPN, 2) determine structural and functional brain correlates of painful CIPN in the DPMN in NHBs and NHWs, and 3) determine inflammatory mediators in patients with painful CIPN and their relationship to the severity of painful CIPN and DPMN structure and function. The investigators expect NHB subjects will experience greater therapeutic effects of tDCS compared to NHW subjects, since NHBs have a dysregulated DPMN potentially affected by neuroinflammation. The goals of this project align with the mission of RCMI@Morgan to understand and combat urban health disparity issues in the City of Baltimore and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, and comprehend English
* Non-Hispanic White or Non-Hispanic Black
* Stable medication dosage over previous 4 weeks
* Completed primary surgery or chemotherapy for cancer at least 3 months prior to signing consent form
* Diagnosed with painful chemotherapy-induced neuropathy

Exclusion Criteria:

* Chronic pain due to another painful condition (e.g., fibromyalgia, chronic low back pain, etc.)
* Any neurological deficits (e.g., lower extremity weakness or bowel/bladder dysfunction, etc.)
* Deficient folate levels (<7 nmol/ml serum)
* Deficient vitamin B12 levels (<200 pg/mL serum)
* Deficient Vitamin D levels (<50 nmol/L or <20 ng/ml)
* Comorbidities affecting sensorimotor function (e.g., multiple sclerosis, diabetes, etc.)
* Unstable mental health condition (acute medical management/hospitalization in the past 6 mo.)
* Elevated hemoglobin A1c levels indicative of uncontrolled diabetes (>6.5%)
* Self-reported Substance abuse (current)
* Drug test positive for illicit drugs except THC
* Excessive alcohol consumption defined as: 1) More than 3 glasses of wine a day; 2) More than 3 beers a day; 3) More than 60 mL of hard liquor a day
* Presence of cardiac pacemaker or automatic implantable cardioverter-defibrillator (AICD).
* Pregnancy, lactation (will be screened with urine pregnancy test)
* Non-removable metal or tattoos around head, excepting dental appliances and fillings
* Use of implantable copper birth control device
* History of frequent severe headaches
* Unstable coronary artery disease
* Uncontrolled Seizure disorder
* Uncontrolled hypertension
* Stage IV cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants able to adhere to the at home remote stimulation protocol | 2 weeks
  Number of participants able to adhere to the at home study protocol comparing non-Hispanic blacks to non-Hispanic whites for both active and sham stimulation groups
Number of side effects reported on the transcranial direct current stimulation side effect questionnaire | 2 weeks
  Number of side effects reported on the transcranial direct current stimulation side effect questionnaire comparing non-Hispanic blacks to non-Hispanic whites for both active and sham stimulation groups (n=20 per group; 4 groups)
Cortical thickness | 10 minutes
  Cortical thickness comparison between non-Hispanic blacks and non-Hispanic whites
Blood oxygen level dependent (BOLD) response to sharp mechanical stimuli | 10 minutes
  Comparison between non-Hispanic black and non-Hispanic white participants with and without painful chemotherapy induced peripheral neuropathy
Blood oxygen level dependent (BOLD) response to painful heat stimuli | 10 minutes
  Comparison between non-Hispanic black and non-Hispanic white participants with and without painful chemotherapy induced peripheral neuropathy
Blood oxygen level dependent (BOLD) response to cold heat stimuli | 10 minutes
  Comparison between non-Hispanic black and non-Hispanic white participants with and without painful chemotherapy induced peripheral neuropathy

SECONDARY OUTCOMES:
Brief pain inventory short form score | 2 weeks
  Comparing active to sham transcranial direct current stimulation in non-Hispanic black participants and non-Hispanic white participants
Brief pain inventory short form score | At 6 week follow-up
  Comparing active to sham transcranial direct current stimulation in non-Hispanic black participants and non-Hispanic white participants

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cynthia Renn, Baltimore, Maryland
  - Morgan State University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be shared through supplementary materials in primary journals and by 01/2030 are planned to be shared in data repositories or journals.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Study protocol and statistical analysis plan are planned to be submitted to a per-registration service or journal about December 2024.
  Clinical study reports and structural and functional MRI will be submitted to data repositories or peer-reviewed data journals and the Enhancing Neuro Imaging Genetics through Meta Analysis (ENIGMA) Chronic Pain Working group by about December 2030.
Access Criteria: Any de-identified data not published will be available from the study authors upon reasonable request.